CLINICAL TRIAL: NCT07399873
Title: Outcomes From Point-of-Care STI Testing in an Urban Sexual Health Clinic: A Randomized Trial
Brief Title: Outcomes From Point-of-Care Sexually Transmitted Infection (STI) Testing in an Urban Sexual Health Clinic: A Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Roche Diagnostic Ltd. (Industry)
Responsible Party: Principal Investigator, Kevin L, Ard, Director, Sexual Health Clinic, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2025P002645
Record Dates: First submitted 2026-01-04; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neisseria Gonorrhoeae Infection; Chlamydia Trachomatis Infection
Keywords: gonorrhea; chlamydia; sexually transmitted infection; STI; point-of-care testing
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (Active Comparator): Participants randomized to the standard-of-care arm will receive STI testing via a routine, laboratory-based assay for C. trachomatis and N. gonorrhoeae.
  Interventions: Diagnostic Test: Laboratory-based chlamydia and gonorrhea NAAT
- Point-of-care Testing (Experimental): Participants randomized to this arm will receive a point-of-care testing in addition to standard, laboratory-based testing for C. trachomatis and N. gonorrhoeae.
  Interventions: Diagnostic Test: Point-of-care assay for chlamydia and gonorrhea; Diagnostic Test: Laboratory-based chlamydia and gonorrhea NAAT
- CRISPR-based Assay Assessment (Other): Participants in this arm will have collection of additional samples for testing via a research-only, novel CRISPR-based assay for STIs and antimicrobial resistance.
  Interventions: Diagnostic Test: CRISPR-based assay

INTERVENTIONS:
Diagnostic Test: Point-of-care assay for chlamydia and gonorrhea — This intervention consists of use of Cobas® Liat CT/NG Assay (Roche, United States).
  Arms: Point-of-care Testing
Diagnostic Test: Laboratory-based chlamydia and gonorrhea NAAT — This intervention consists of routine, laboratory-based diagnostic testing for chlamydia and gonorrhea via nucleic acid amplification.
  Arms: Point-of-care Testing; Standard of Care
Diagnostic Test: CRISPR-based assay — This is a novel assay using CRISPR technology to assess for STIs and antimicrobial resistance.
  Arms: CRISPR-based Assay Assessment

SUMMARY:
The goal of this clinical trial is to learn about the impact of a point-of-care test for gonorrhea and chlamydia in people without symptoms who are seeking sexually transmitted infection testing. The main questions it aims to answer are:

Does the point of care test reduce the time to antibiotic treatment? Does the point of care test increase the number of people who have completed treatment by day 7?

Researchers will compare the point-of-care test to a standard laboratory-based test for gonorrhea and chlamydia.

Participants will be asked to provide a urine sample or vaginal swab for testing. They will also complete surveys about their experiences with the testing.

DETAILED DESCRIPTION:
Investigators will prospectively enroll asymptomatic individuals presenting for STI screening. Individuals will be randomized in a 1:1 manner to receive either standard-of-care screening or standard-of-care plus point-of-care testing for Chlamydia trachomatis and Neisseria gonorrhoeae. Among individuals enrolled and randomized to the intervention arm, investigators will collect an additional vaginal swab among women or urine sample among men for point-of-care testing using the Cobas® Liat CT/NG Assay (Roche, United States). Individuals who test positive for either pathogen (in either arm) will receive treatment according to Centers for Disease Control and Prevention (CDC) guidelines. The time to treatment and the proportion of patients who are on or have completed treatment at day 7 day after the initial visit will be evaluated.

Primary Objective: To compare the time to antimicrobial therapy initiation for C. trachomatis and/or N. gonorrhoeae among patients treated according to a point-of-care test plus standard of care versus patients treated according to standard of care alone.

Secondary Objective: To evaluate the proportion of patients who have completed or have started therapy by day 7 after a positive C. trachomatis and/or N. gonorrhoeae test result among patients treated according to a point-of-care test plus standard of care versus patients treated according to standard of care alone.

As a second aim, investigators will seek to compare performance of a novel clustered regularly interspaced short palindromic repeats (CRISPR)-based point-of-care STI and antimicrobial resistance assay to reference testing on additional samples collected from symptomatic participants in this study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Willing and able to provide informed consent
* Asymptomatic at the urogenital site
* Being screened for urogenital C. trachomatis and/or N. gonorrhoeae as part of routine clinical care

Exclusion Criteria:

* Indication for antimicrobial therapy for C. trachomatis or N. gonorrhoeae at the time of the visit, regardless of test results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Days to antibiotic initiation | Time in days (0-365)
  Time, in days, to initiation of antimicrobial therapy for C. trachomatis and N. gonorrhoeae

SECONDARY OUTCOMES:
Antimicrobial therapy initiation within 7 days | 7 days from baseline
  Number and proportion of patients completing or starting antimicrobial therapy by day 7 after a positive test for C. trachomatis or N. gonorrhoeae

OTHER OUTCOMES:
CRISPR-based assay performance | At baseline
  Comparison of performance of the CRISPR-based assay to reference testing as measured by the sensitivity and specificity of the CRISPR-based assay for detection Chlamydia trachomatis and Neisseria gonorrhoeae, in relationship to reference testing.

IPD SHARING:
Plan to Share IPD: Yes
We will share the de-identified data, study protocol, and analysis plan no later than the time of publication for a period of 2 years.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: We plan to share this information beginning no later than the time of publication for a period of 2 years.
Access Criteria: Researchers will be able to access the information upon request from the investigators, with a description of what the researchers propose to do with the data. A data sharing agreement must be established and approved by both parties' institutions for data sharing to take place. Requests for data sharing will be reviewed by the principal investigator and co-investigator.